CLINICAL TRIAL: NCT04514419
Title: A Phase III Study to Compare HS627 vs. Pertuzumab on the Efficacy, Safety and Immunogenicity in Combination With Trastuzumab and Docetaxel as Neoadjuvant Therapy in Patients With Early-stage or Locally Advanced HER2 Positive Breast Cancer
Brief Title: Treatment of Breast Cancer With Trastuzumab + HS627/ Pertuzumab + Docetaxel
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioRay Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS627-III
Record Dates: First submitted 2020-07-30; First posted 2020-08-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Docetaxel; pertuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trastuzumab + HS627 + Docetaxel (Experimental): Trastuzumab HS627 Docetaxel
  Interventions: Drug: HS627
- Trastuzumab + Pertuzumab + Docetaxel (Experimental): Trastuzumab Pertuzumab Docetaxel
  Interventions: Drug: Pertuzumab

INTERVENTIONS:
Drug: HS627 — Prior to surgery: trastuzumab, HS627, and docetaxel for 4 cycles (1 cycle = 21 days).
  Other Names: Trastuzumab + HS627 + Docetaxel
  Arms: Trastuzumab + HS627 + Docetaxel
Drug: Pertuzumab — Prior to surgery: trastuzumab, Pertuzumab, and docetaxel for 4 cycles (1 cycle = 21 days).
  Other Names: Trastuzumab Pertuzumab Docetaxel
  Arms: Trastuzumab + Pertuzumab + Docetaxel

SUMMARY:
The trial included screening period (4 weeks) and treatment period (4 treatment cycles, at least 12 weeks).

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, positive drug parallel control design was used. The trial included screening period (4 weeks) and treatment period (4 treatment cycles, at least 12 weeks). All eligible subjects were randomly divided into experimental group (hs627 treatment group) and control group (pertuzumab) treatment group. After 4 treatment cycles, the subjects arranged surgical treatment, and then conducted the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast carcinoma with a primary tumor size of more than (>) 2 centimeters (cm) by standard local assessment technique；
* Breast cancer stage at presentation: early-stage (T2-3, N0-1, M0), locally advanced (T2-3, N2-3,M0 or T4a-c, any N, M0), or infl ammatory (T4d, any N,M0)；
* Known hormone receptor status (estrogen receptor and/or progesterone receptor)；
* HER2 positive (HER2+++ by IHC or ISH+).
* Baseline left ventricular ejection fracture >= 55% measured by echocardiography (preferred) or multiple gated acquisition scan；
* Normalities in liver, kidney or hematologic function laboratory tests immediately prior to randomization;
* Absolute value of neutrophils ≥ 1.5 × 109 / L;
* Platelet ≥ 90×109 / L;
* Hemoglobin ≥ 90g / L;
* Serum creatinine≤ 1.5 times the upper limit of normal (ULN);
* Serum total bilirubin≤1.5 times ULN (except for Gilbert syndrome);
* Aspartate aminotransferase (AST) and / or alanine aminotransferase (ALT) ≤ 1.5-fold ULN;
* International normalized ratio (INR), activated partial prothrombin time (APTT) ≤ 1.5 times ULN.
* ECOG≤1；

Exclusion Criteria:

* Stage IV metastatic ;
* Bilateral breast cancer;
* Previous anti-cancer therapy or radiotherapy for any malignancy;
* History of other malignancy within 5 years, except for appropriately-treated carcinoma in Cervical carcinoma in situ, basal cell carcinoma or squamous cell skin cancer;
* Serious cardiac illness or medical condition;
* HIV antibody positive; HCV antibody positive and HCV RNA positive; HBcAb or HBsAg positive, and HBV DNA positive;
* Sensitivity to any of the study medications, any of the ingredients or excipients of these medications;
* Known mental history had poor compliance;
* Known to have drug abusers;
* Concurrent anti-cancer treatment in another investigational trial, including hormone therapy, bisphosphonate therapy, or immunotherapy;
* Needed intravenous antibiotic treatment due to infection within 7 days before random enrollment;
* Major surgical procedure unrelated to breast cancer within 4 weeks prior to randomization or expected to perform major surgery during the trial period;
* Premenopausal women (menopause is defined as non treatment induced menopause≥12 months) or without surgical sterilization (e.g., ovariectomy and / or uterus): refuse to take one or more effective contraceptive measures during treatment and at least 6 months after the last study treatment; blood pregnancy test is positive; pregnant or lactating women; Considered unsuitable for the study or may not be able to complete the trial due to other reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2020-06-28 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving Pathological Complete Response (pCR) as Assessed by the Independent Review Committee (IRC) | After surgery (At surgery cycle 4 Days 22-35)(1 cycle = 21 days)
  pCR was defined as ypT0/is According to the American Joint Committee on Cancer Staging System as Assessed by the IRC

SECONDARY OUTCOMES:
Percentage of Participants With Total Pathologic Complete Response (tpCR) as Assessed by the Independent Review Committee (IRC) | After surgery (At surgery cycle 4 Days 22-35) (1 cycle = 21 days)
  tpCR was defined as ypT0/is, ypN0 as assessed by an Independent Review Committee (IRC)
Percentage of Participants With pCR as Assessed by the Local Pathologist | After surgery (At surgery cycle 4 Days 22-35) (1 cycle = 21 days)
  pCR was defined as ypT0/is as assessed by Local Pathologist
Percentage of Participants With Total Pathologic Complete Response (tpCR) as Assessed by the Local Pathologist | After surgery (At surgery cycle 4 Days 22-35) (1 cycle = 21 days)
  tpCR was defined as ypT0/is, ypN0 as assessed by Local Pathologist
Percentage of Participants With an Objective Response | Prior to surgery (Cycle 4 Days 21) (1 cycle = 21 days)
  An objective response was defined as the percentage of participants who achieved a complete response or partial response as the best tumor response during the treatment period (that is, during Cycles 1-4 prior to surgery), as determined by the investigator on the basis of Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Percentage of Participants with vital signs, physical examination, left ventricular ejection fraction (LVEF), laboratory examination, adverse events (AE) until last visit | Last Visit （After surgery 8 days）（After 4 cycles treatment ，After surgery ） (1 cycle = 21 days)
  The percentage of participants who experienced at least one vital sign, physical examination, left ventricular ejection fraction (LVEF), laboratory examination, adverse events (AE) during the study is reported here.

CONTACTS AND LOCATIONS:
Overall Officials: Zefei Jiang, M.D, Principal Investigator — The Affiliated Hospital of Qingdao University; Haibo Wang, M.D, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China